CLINICAL TRIAL: NCT03236675
Title: Detection of Either the EML4-ALK Gene Rearrangements or the T790M EGFR Mutation in the Plasma of Advanced NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2015-003A
Record Dates: First submitted 2016-02-24; First posted 2017-08-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10-20 mL of whole blood collected in K2EDTA Plasma Preparation Tubes (PPT) will be acquired via standard venipuncture.
  This will be an observational study as subjects will only provide plasma specimens at different time points and no therapeutic or intervention will be received outside of their normal standard of care.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EML4-ALK: ALK positive patients
- T790M EGFR: T790M positive patients

SUMMARY:
Demonstrate feasibility of detection of EML4-ALK fusion transcripts and T790M EGFR mutation from exosomes in the circulation of Non-Small Cell Lung Cancer (NSCLS) patients.

DETAILED DESCRIPTION:
The goal of this study is two-fold: 1) Demonstrate feasibility of detection of EML4-ALK fusion transcripts in the circulation of NSCLC patients positive for ALK on tissue analysis, using an institutionally accepted assay; 2) Demonstrate feasibility of detection of T790M EGFR mutation in the circulation of NSCLC patients positive for T790M on tissue analysis, using an institutionally accepted assay.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed NSCLC, stage IIIB- IV, and have tested positive for the presence of EML4-ALK on tissue specimen, fresh or archived, using an institutionally accepted assay.
2. Age of 18 years or older.
3. Participants are being considered for ALK-directed therapy or have progressed on EGFR TKI treatment.
4. Participants must have hemoglobin > 10 mg/dL.
5. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Hepatitis (all types) in patient's medical record
2. HIV documented in patient's medical record
3. Hemoglobin < 10 mg/dL
4. Less than 18 years of age
5. Histologically confirmed NSCLC Stage I-IIIA
6. Tested negative for the presence of EML4-ALK and T790M EGFR on tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
ALK mutation by tissue assay. | Two years
  Patients found to be positive for ALK mutation by tissue assay. ALK fusions in samples will be considered binary - positive or negative/ not assessable. 2x2 table will be constructed to determine concordance with tissue testing.
T790M EGFR mutation by tissue assay | Two years
  Patients found to be positive for T790M EGFR mutation by tissue assay. ALK fusions in samples will be considered binary - positive or negative/ not assessable. 2x2 table will be constructed to determine concordance with tissue testing.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Tun, Study Director — Exosome Diagnostics, Inc.
Locations (2):
- United States (2):
  - Memorial Healthcare System, Hollywood, Florida
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided